CLINICAL TRIAL: NCT01500148
Title: Clinical Assessment of the St. Jude Medical (SJM) Percutaneous Mitral Valve Repair (PMVr) Device Concept
Brief Title: St. Jude Medical Percutaneous Mitral Valve Repair Study
Acronym: SJM PMVr
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1101
Record Dates: First submitted 2011-12-06; First posted 2011-12-28 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Mitral Valve Prolapse
Keywords: Mitral Valve Prolapse; Mitral Valve Disease; Mitral Valve Regurgitation; Mitral Valve Insufficiency; Mitral Valve Incompetence; Percutaneous Mitral Valve Repair; Posterior leaflet prolapse; Mitral valve degeneration
MeSH Terms: conditions — Mitral Valve Prolapse; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intevention-PMVr Procedure (Experimental)
  Interventions: Device: PMVr procedure (SJM Percutaneous Mitral Valve Repair (PMVr)

INTERVENTIONS:
Device: PMVr procedure (SJM Percutaneous Mitral Valve Repair (PMVr) — A maximum of ten (10) subjects will receive a percutaneous mitral valve clip procedure.

SUMMARY:
The purpose of this proof-of-concept study is to assess the relative safety and feasibility of the SJM Percutaneous Mitral Valve Repair (PMVr) Device.

DETAILED DESCRIPTION:
Subjects will be followed-up through 6 weeks post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has symptomatic or asymptomatic moderate (2+) or severe (3-4+) mitral regurgitation.
* Subject has an ejection fraction (EF) ≥ 30%.
* Subject is of legal age (≥18 years old).
* Subject is planned to undergo surgical repair or replacement of the mitral valve for symptomatic or asymptomatic posterior leaflet mitral prolapse.

Exclusion Criteria:

* Subject requires a complex mitral valve repair or has isolated anterior prolapse.
* Subject has mitral valve stenosis in which the annulus opening is <10mm. Subject has valve disease other than mitral which requires surgical intervention.
* Subject requires a concomitant procedure.
* Subject has a pre-existing prosthetic valve in any position.
* Subject had stenting or PCI within 6 months before the planned procedure, or is anticipated to require stenting or PCI within 6 months post-procedure.
* Subject has calcification of the mitral leaflets or annulus which in the medical opinion of the surgical investigator would limit repair and /or implantation of the investigational device.
* Subject has renal insufficiency or is on chronic dialysis.
* Subject has had a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months.
* Subject has a history of endocarditis or has active endocarditis.
* Subject has a history of autoimmune disease.
* Subject has significant known carotid artery disease.
* Subject has an aorto-mitral angle of <110 degrees.
* Subject has hypertrophic obstructive cardiomyopathy (HOCM's Disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Device and Procedural Success | During the investigational procedure
  The primary objective is to evaluate the technical feasibility and acute device deployment characteristics of the SJM PMVr Device.
  Technical feasibility and deployment characteristics will be defined as:
  * The ability of the delivery system to access the mitral valve
  * The ability of the device to capture mitral valve (MV) leaflet tissue
  * Ability to plicate MV leaflet tissue
  * The clip is able to be deployed in MV leaflet tissue
  * The delivery system is able to be removed.

SECONDARY OUTCOMES:
Quantification of SAEs reported that are unique to the investigational procedure | Through 6 weeks post-implantation
  The secondary objective is to evaluate safety of the SJM PMVr device by summarizing SAEs unique to accessing the valve, placing the clip, and removing the delivery system.

CONTACTS AND LOCATIONS:
Locations (1):
- Papworth Hospital, Cambridge, United Kingdom